CLINICAL TRIAL: NCT00515359
Title: RCT for Intermittent Versus Continuous Propofol Sedation for Pediatric Brain and Spine MRI Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Helen DeVos Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-140
Record Dates: First submitted 2007-08-07; First posted 2007-08-13 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Encephalopathy; Developmental Delay and Behavioral Changes; Cord Tumor Compression or Instability; Cord Tethering or Malformation
Keywords: Sedation; MRI; pediatric; propofol; brain; spine; quality of MRI; Continuous propofol dosing; continuous propofol administration; Intermittent propofol dosing; intermittent propofol administration; Sedative agent; propofol continuous infusions; Recovery time; Complications of sedation; bolus dosing
MeSH Terms: conditions — Brain Diseases; Learning Disabilities; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Dosing (Active Comparator): continuous dosing
  Interventions: Procedure: Continuous Propofol Sedation
- Intermittent Dosing (Active Comparator): Intermittent Dosing
  Interventions: Procedure: Intermittent Propofol Sedation

INTERVENTIONS:
Procedure: Intermittent Propofol Sedation — Intermittent versus continuous dosage
  Arms: Intermittent Dosing
Procedure: Continuous Propofol Sedation — intermittent vs continuous dosage
  Arms: Continuous Dosing

SUMMARY:
RCT for Intermittent versus Continuous Propofol Sedation for Pediatric Brain and Spine MRI Studies

DETAILED DESCRIPTION:
A study comparing the dose of propofol used as a continuous infusion versus intermittent bolus dosing looking at recovery time complications, and quality of the MRI studies in Pediatric Sedation Services for patients age 1 month to 18 years receiving an brain or spine MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month to 18 years
* Receiving a brain or spine MRI with propofol sedation
* Deemed safe to undergo sedation with propofol based on a pre-sedation examination
* Patient judged not to require any pre-medication with any other medication except nasal decongestants or anticholinergic medications

Exclusion Criteria:

* Patient below or above set age limits.
* Patient requires MRI studies on other body areas.
* Patient requires pre-medication with a sedative or tranquilizer
* Patient requires additional medications during sedation to complete the procedure.
* Propofol is being used as a rescue sedative to complete the procedure.
* Propofol is being used as a rescue sedative to complete a procedure that was initiated by another sedative.
* Patients who develop complications that require termination of the imaging procedure will not be included in the dose or recovery time calculations, but the complication will be counted as such in their respective group and study will be reported as non-diagnostic.
* Insulin dependent diabetes
* Thyroid disease

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 276 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
to compare recovery time, complications and quality of the MRI studies when continuous infusion of propofol was used versus intermittent bolus dosing | study completion

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Hassan, MD, Principal Investigator — Helen DeVos Children's Hospital
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

REFERENCES:
- See also: Spectrum Health — https://corewellhealth.org/